CLINICAL TRIAL: NCT04040751
Title: Carepartner Collaborative Integrated Therapy in Sub-Acute Stroke
Acronym: CARE-CITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sarah Blanton, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00107906; R21NR018015 (NIH)
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Stroke
Keywords: Telehealth; Rehabilitation; Care partner; Sub-acute stroke; CARE-CITE; Stroke survivors
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CARE-CITE Carepartner (Experimental): This study arm consists of carepartners receiving the CARE-CITE intervention. The CARE-CITE intervention will occur over 4 weeks in the dyad's home. The research interventionist will conduct two in-home visits (at orientation and during week 4), two phone call visits (at weeks 2 and 3), and one telephone follow up at week 8.
  Interventions: Behavioral: CARE-CITE
- Control Carepartners (Active Comparator): Carepartners in this study arm receive customary care outpatient rehabilitation therapy but no CARE-CITE intervention. The carepartner will receive the same number of structured weekly phone calls and the "booster call" to answer any questions, assess helpfulness of the information and ascertain if there was any use of the web resources or social support groups.
  Interventions: Behavioral: Standard of care
- CARE-CITE Stroke Survivor (Experimental): This study arm consists of stroke survivors of carepartners receiving the CARE-CITE intervention. The CARE-CITE intervention will occur over 4 weeks in the dyad's home. The research interventionist will conduct two in-home visits (at orientation and during week 4), two phone call visits (at weeks 2 and 3), and one telephone follow up at week 8.
  Interventions: Behavioral: CARE-CITE
- Control Stroke Survivors (Active Comparator): Stroke survivors in this study arm receive customary care outpatient rehabilitation therapy but no CARE-CITE intervention. Carepartners of the stroke survivors will receive the same number of structured weekly phone calls and the "booster call" to answer any questions, assess helpfulness of the information and ascertain if there was any use of the web resources or social support groups.
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: CARE-CITE — The primary CARE-CITE components will be education via web platform. Carepartners complete 6 online CARE-CITE modules (15-30-minute sessions each). The modules include demonstration videos and instructive content covering following areas: principles of functional task practice (i.e., activities of daily living such as eating, grooming, or leisure/vocational activities), adaptation of tasks, and importance of progression of challenging tasks to drive neuroplasticity (i.e., increasing numbers of practice repetitions or weight of objects lifted). Underpinning the content is the concept of autonomy support, with examples of fostering empathy, problem solving, instruction in the use of non-controlling language with role playing situations and the importance of creating choice in activities.
  Arms: CARE-CITE Carepartner; CARE-CITE Stroke Survivor
Behavioral: Standard of care — The carepartner will receive a support brochure with general caregiving information including website resources to mimic web interaction of intervention group (e.g., stroke caregiver resource site).
  Arms: Control Carepartners; Control Stroke Survivors

SUMMARY:
Carepartner and Collaborative Integrated Therapy (CARE-CITE) is a novel, web-based carepartner focused intervention designed to foster problem solving and skill building while facilitating carepartner engagement during upper extremity functional activities in the home setting. The proposed study will evaluate the application of the CARE-CITE intervention paired with usual and customary care during the sub-acute stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of serious, long-term disability in the United States, and has a particularly harmful impact on individuals and families. Approximately 4.8 million stroke survivors require assistance from family members who are often untrained and ill prepared for the burdens associated with stroke rehabilitation. Family carepartners are key contributors to stroke recovery, but their efforts can lead them to experience a high level of burden and depressive symptoms, reduced quality of life and increased stress in the context of high levels of family conflict surrounding the recovery process. Rehabilitation therapy interventions have primarily targeted stroke survivor outcomes without specifically addressing the well-being of the carepartner.

The researchers of this study have developed a theory-based, family-centered intervention, Carepartner and Collaborative Integrated Therapy (CARE-CITE), designed to engage carepartners during stroke survivor upper extremity (UE) functional task practice in the home. Residual UE impairments occur in up to 80% of stroke survivors and are a primary factor in loss of functional independence. CARE-CITE guides the carepartner in collaborative goal setting and providing autonomy support (characterized by empathy, choice and reducing use of controlling language) for the stroke survivor to promote motivation and creative problem solving in UE self-management.

Participating stroke survivor and carepartner dyads will be randomized to receive the CARE-CITE intervention with usual customary care, or usual customary care alone for four weeks.

ELIGIBILITY:
Inclusion Criteria for Stroke Survivors:

* 1-3 months post ischemic or hemorrhagic event
* discharged from inpatient neurologic rehabilitation to their home
* have minimal to moderate upper extremity (UE) deficits (actively initiate 20 degrees of wrist and 10 degrees of finger extension)
* no severe cognitive deficits (Mini -mental test >24)
* no physician determined major medical problems that would limit participation in outpatient therapy

Inclusion Criteria for Carepartners:

* spouse/partner or family member
* dwelling in the same household
* self-identify as the primary caregiver of the stroke survivor
* >21 years old
* able to read and write English
* have no significant cognitive deficits (Mini -mental test >24)
* familiar with using a computer and accessing websites, or with using a tablet

Exclusion Criteria:

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Blanton, PT, DPT, Principal Investigator — Emory University
Locations (1):
- Emory Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, will be shared after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following final publication of the results of the aims.
Access Criteria: Researchers who provide a methodologically sound proposal and whose proposed use of data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Proposals should be directed to sarah.blanton@emory.edu. To gain access, data requestors will need to sign a data access agreement. The data agreement will be reviewed by the investigative team for approval.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began August 9, 2019 and all follow up was complete by December 21, 2021. Participants were enrolled from Emory Hospital in Atlanta, Georgia, USA.
Groups:
- Control Carepartners: Carepartners receiving customary care outpatient rehabilitation therapy but no CARE-CITE intervention. The carepartner will receive the same number of structured weekly phone calls and the "booster call" to answer any questions, assess helpfulness of the information and ascertain if there was any use of the web resources or social support groups.
- Control Stroke Survivors: Stroke survivors receiving customary care outpatient rehabilitation therapy but no CARE-CITE intervention. The carepartner of the stroke survivor will receive the same number of structured weekly phone calls and the "booster call" to answer any questions, assess helpfulness of the information and ascertain if there was any use of the web resources or social support groups.
Period: Overall Study
Arm/Group | CARE-CITE Carepartner | Control Carepartners | CARE-CITE Stroke Survivor | Control Stroke Survivors
Started | 17 | 6 | 17 | 6
Completed | 15 | 6 | 15 | 6
Not Completed | 2 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- CARE-CITE Carepartner: Carepartners receiving the CARE-CITE intervention
- Control Carepartners: Carepartners receiving customary care outpatient rehabilitation therapy but no CARE-CITE intervention
- CARE-CITE Stroke Survivor: Stroke survivors of carepartners receiving the CARE-CITE intervention
- Control Stroke Survivors: Stroke survivors receiving customary care outpatient rehabilitation therapy but no CARE-CITE intervention
- Total: Total of all reporting groups
Arm/Group | CARE-CITE Carepartner | Control Carepartners | CARE-CITE Stroke Survivor | Control Stroke Survivors | Total
Number analyzed (Participants) | 17 | 6 | 17 | 6 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.6) | 58.5 (12.2) | 60.6 (11.4) | 60.7 (13.4) | 58.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 9 | 2 | 29
  Male | 4 | 1 | 8 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Asian | 2 | 0 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 0 | 8 | 1 | 17
  White | 6 | 5 | 5 | 4 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 6 | 17 | 6 | 46
Education [Count of Participants; unit: Participants]
  High school or less | 3 | 0 | 4 | 0 | 7
  1-3 years of college | 3 | 3 | 3 | 4 | 13
  4 or more years of college | 11 | 3 | 10 | 2 | 26

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiologic Studies - Depression (CES-D) Scale Score Among Carepartners
Description: Depression among carepartners was assessed with the CES-D. The CES-D is 20-item, 4-point Likert-type scale where 0 = none/rare and 3 = most or all of the time. The scoring of positive items is reversed. The possible range of scores is 0 to 60, with the higher scores indicating the presence of more symptomatology. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Carepartner | Control Carepartners
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 9.9 (9.7) | 11.2 (8.5)
  2 Months Post-intervention | 9.1 (8.2) | 9.3 (4.8)

2. Primary Outcome: Short Form Health Survey (SF-36) Scale Score Among Carepartners
Description: Carepartner quality of life was assessed with the SF-36. The SF-36 is a 36-item Likert-type scale, mental health domain. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. Lower scores indicate greater disability, while higher scores indicate less disability (i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability). Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Carepartner | Control Carepartners
Number analyzed (Participants) | 17 | 6
score on a scale
  Physical Functioning - Baseline | 73.9 (21.6) | 92.5 (8.2)
  Physical Functioning - 2 Months Post-intervention | 82.3 (13.1) | 85.8 (15.6)
  Role Limitation, Physical - Baseline | 70.6 (42.6) | 83.3 (20.4)
  Role Limitation, Physical - 2 Months Post-intervention | 76.7 (38.3) | 70.8 (45.9)
  Role Limitation, Emotional - Baseline | 70.6 (30.4) | 91.7 (13.9)
  Role Limitation, Emotional - 2 Months Post-intervention | 82.2 (18.3) | 83.3 (14.9)
  Energy/Vitality - Baseline | 58.2 (21.1) | 47.5 (27.2)
  Energy/Vitality - 2 Months Post-intervention | 64.0 (16.4) | 55.0 (28.1)
  Emotional Well Being - Baseline | 74.6 (18.9) | 74.0 (12.3)
  Emotional Well Being - 2 Months Post-intervention | 76.3 (16.0) | 81.3 (12.8)
  Social Functioning - Baseline | 76.5 (22.5) | 83.3 (30.3)
  Social Functioning - 2 Months Post-intervention | 83.3 (23.5) | 83.3 (21.9)
  Pain - Baseline | 81.0 (16.8) | 78.8 (13.9)
  Pain - 2 Months Post-intervention | 77.2 (22.6) | 73.8 (31.7)
  General Health - Baseline | 67.4 (10.5) | 72.5 (7.6)
  General Health - 2 Months Post-intervention | 71.0 (9.7) | 76.7 (5.2)

3. Primary Outcome: Wolf Motor Function Test (WMFT) Upper Extremity Function Ability Score (FAS)
Description: The Wolf Motor Function Test (WMFT) assesses upper extremity motor ability with 17 timed and functional tasks (15 timed and 2 strength tasks). Functional ability for each task is scored from 0 to 5, where 0 = does not attempt with upper extremity being tested, and 5 = movement appears to be normal. Total scores range from 0 to 85 and lower scores indicate lower functional ability. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Population: The WMFT is an in-person assessment and administration of the WMFT was stopped after the study converted to fully remote delivery due to Coronavirus Disease 2019 (COVID-19) pandemic health restrictions which limited in-person visits. This analysis includes participants who completed the WMFT assessment prior to the study being conducted remotely.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Stroke Survivor | Control Stroke Survivors
Number analyzed (Participants) | 5 | 2
score on a scale
  Baseline | 59.0 (3.9) | 43.0 (5.7)
  2 Months Post-intervention: number analyzed (Participants) | 2 | 2
  2 Months Post-intervention | 59.5 (7.8) | 55.5 (0.7)

4. Primary Outcome: Wolf Motor Function Test (WMFT) Test Time Among Stroke Survivors
Description: The Wolf Motor Function Test (WMFT) assesses upper extremity motor ability with 17 functional tasks (15 timed and 2 strength tasks). The time, in seconds, required to complete each of 15 timed scores is calculated, with lower times (faster speeds) indicating higher functioning levels. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | CARE-CITE Stroke Survivor | Control Stroke Survivors
Number analyzed (Participants) | 5 | 2
seconds
  Baseline | 4.2 (3.9) | 27.9 (34.4)
  2 Months Post-intervention: number analyzed (Participants) | 2 | 2
  2 Months Post-intervention | 2.8 (0.3) | 2.7 (0.8)

5. Primary Outcome: Quality of Upper Extremity Function by Motor Activity Log (MAL) Score Among Stroke Survivors
Description: The Motor Activity Log is 30-item questionnaire assessing use of the affected arm during normal daily activities. Responses are given on a Likert scale where 0 = the weaker arm was not used at all for that activity (never) to 5 = the ability to use the weaker arm for that activity was as good as before the stroke (normal). The total score is the average of all items and ranges from 0 to 5, where higher values indicate greater function of the arm that was impacted by the stroke. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Population: This analysis includes participants who completed both the Baseline and 2 Months Post-intervention assessment. One dyad in the CARE-CITE study arm withdrew from the study after completing some of the questionnaires of the 2 Months-Post intervention evaluation but did not complete the remote assessment in which the MAL was administered.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Stroke Survivor | Control Stroke Survivors
Number analyzed (Participants) | 16 | 6
score on a scale
  Baseline | 2.4 (1.3) | 2.2 (1.1)
  2 Months Post-intervention | 3.4 (1.0) | 3.3 (1.2)

6. Primary Outcome: Stroke Impact Scale (SIS) Score Among Stroke Survivors
Description: Quality of life among stroke survivors was assessed with the Stroke Impact Scale (SIS). The SIS is a stroke specific, self report questionnaire (59 items across 8 domains) that measures how a stroke has impacted a participant's health and life, including strength, memory and thinking, emotions and mood, communication, activities of daily living, mobility, function of affected upper extremity, and social participation. Each item is rated in a 5-point Likert scale in terms of the difficulty the participant has experienced in completing each item. A score for each domain is obtained, ranging from 0 to 100 where higher scores indicate greater ability to perform tasks. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Stroke Survivor | Control Stroke Survivors
Number analyzed (Participants) | 17 | 6
score on a scale
  Strength Domain Score - Baseline | 50.4 (21.7) | 56.3 (10.5)
  Strength Domain Score - 2 Months Post-Intervention | 64.2 (19.5) | 58.3 (10.9)
  Memory and Thinking Domain Score - Baseline | 76.3 (28.5) | 73.8 (16.1)
  Memory and Thinking Domain Score - 2 Months Post-Intervention | 91.7 (12.0) | 82.7 (22.2)
  Emotions and Mood Domain Score - Baseline | 60.0 (10.7) | 61.5 (10.4)
  Emotions and Mood Domain Score - 2 Months Post-Intervention | 60.3 (14.0) | 55.2 (15.4)
  Communication Domain Score - Baseline | 84.9 (27.7) | 76.8 (23.2)
  Communication Domain Score - 2 Months Post-Intervention | 88.8 (18.4) | 78.0 (22.5)
  Activities of Daily Living Domain Score - Baseline | 50.7 (15.3) | 46.7 (14.4)
  Activities of Daily Living Domain Score - 2 Months Post-Intervention | 59.5 (15.7) | 63.7 (10.6)
  Mobility Domain Score - Baseline | 45.9 (23.0) | 57.0 (12.3)
  Mobility Domain Score - 2 Months Post-Intervention | 55.3 (15.3) | 62.2 (16.8)
  Function of Affected Upper Extremity Domain Score - Baseline | 37.4 (22.0) | 25.3 (15.7)
  Function of Affected Upper Extremity Domain Score - 2 Months Post-Intervention | 46.7 (22.0) | 51.3 (27.1)
  Social Participation Domain Score - Baseline | 34.3 (21.1) | 33.3 (26.7)
  Social Participation Domain Score - 2 Months Post-Intervention | 50.0 (18.6) | 32.1 (9.7)

7. Secondary Outcome: Family Care Climate Questionnaire - Carepartners (FCCQ-CP) Score
Description: The Family Care Climate Questionnaire (FCCQ) for carepartners is 14-item questionnaire asking about the carepartners' experiences with the strokes survivor in relation to their rehabilitation activities. Each item is rated on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true). Item scores are averaged to provide an overall score between 1 and 7 where higher scores indicate the carepartner thinks they are providing high autonomy support to the stroke survivor. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Carepartner | Control Carepartners
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 6.3 (0.6) | 6.4 (0.4)
  2 Months Post-intervention | 6.4 (0.3) | 6.6 (0.6)

8. Secondary Outcome: Family Care Climate Questionnaire - Stroke Survivor (FCCQ-SS) Score
Description: The Family Care Climate Questionnaire (FCCQ) for stroke survivors is 14-item questionnaire asking about experiences with family members in relation to rehabilitation activities. Each item is rated on a 7-point Likert scale ranging from 1 (not true at all) to 7 (very true). Item scores are averaged to provide an overall score between 1 and 7 where higher scores indicate the stroke survivor perceives receiving high autonomy support from the carepartner. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Stroke Survivor | Control Stroke Survivors
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 6.6 (0.4) | 6.5 (0.4)
  2 Months Post-intervention | 6.7 (0.4) | 6.3 (1.0)

9. Secondary Outcome: Family Caregiver Conflict Scale (FCCS) Score Among Carepartners
Description: Family conflict was assessed among carepartners with the FCCS. The FCCS is a unidimensional, Likert scale composed of 15 items. For each item, participants indicate their agreement with the item as 1 = not true at all, to 7 = very true. Item scores are summed and total scores range from 15 to 105, where higher scores represent higher levels of conflict within a family. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Carepartner | Control Carepartners
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 21.6 (10.2) | 19.3 (9.7)
  2 Months Post-intervention | 20.9 (8.5) | 20.2 (6.0)

10. Secondary Outcome: Confidence in Hand and Movement Scale (CAHM) Score
Description: Stroke survivor upper extremity self efficacy was assessed with the Confidence in Hand and Movement (CAHM) scale. The CAHM is 20-item instrument where items are scored on a scale of 0 (very uncertain) to 100 (very certain) and averaged to provide a total scale score ranging from 0 to 100. Higher scores indicate greater confidence with performing daily tasks with the impacted arm. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Stroke Survivor | Control Stroke Survivors
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 48.8 (29.2) | 50.5 (28.2)
  2 Months Post-intervention | 67.1 (24.0) | 59.5 (29.9)

11. Secondary Outcome: Family Assessment Device (FAD) Scale Score Among Carepartners
Description: The 12-item General Family Functioning scale from the McMaster Family Assessment Device measures general family functioning. Items are scored on a 4-point scale where 1 = healthy functioning and 4 = unhealthy functioning. A total score is obtained by summing the scores and calculating the average. Higher scores indicate ineffective family functioning. Unadjusted means are presented here.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Carepartner | Control Carepartners
Number analyzed (Participants) | 17 | 6
score on a scale | 1.77 (0.37) | 1.78 (0.33)

12. Secondary Outcome: Caregiver Strain Index (CSI) Score
Description: The CSI is a 13-question tool that measures strain related to care provision. Questions are responded to as either "Yes" or "No" and the total score is determined by summing the "Yes" responses. Total scores range from 0 to 13 and scores of 7 or more indicate high levels of stress. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Carepartner | Control Carepartners
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 4.8 (3.3) | 3.7 (3.3)
  2 Months Post-intervention | 4.5 (3.9) | 4.0 (3.4)

13. Secondary Outcome: Bakas Caregiving Outcomes Scale (BCOS) Score
Description: The BCOS is a unidimensional scale based on 15 items and addresses changes in caregiving social functioning, subjective well-being and physical health. Carepartners respond to statements on a 7-point Likert scale where 1 = changed for the worst, and 7 = changed for the best. Total scores range from 15 - 105 with higher scores representing more positive caregiving outcomes since the stroke. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Carepartner | Control Carepartners
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 57.8 (13.6) | 53.5 (5.8)
  2 Months Post-intervention | 59.9 (8.6) | 55.7 (4.3)

14. Secondary Outcome: Fugl-Meyer Assessment (FMA) Upper Extremity Motor Score
Description: Upper extremity impairment was assessed by the Fugl-Meyer Assessment (FMA). The FMA evaluates and measures recovery in post-stroke hemiplegic patients with 5 domains: motor score (which is further separated for upper and lower extremity), sensation, balance, joint range of motion, and joint pain. Items are scored on a 3-point ordinal scale where 0 = cannot perform and 3 = performs fully. The total score for the upper extremity motor domain ranges from 0 to 66 and a higher score indicates greater arm function. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Population: This analysis includes participants who completed both the Baseline and 2 Months Post-intervention assessment. One dyad in the CARE-CITE study arm withdrew from the study after completing some of the questionnaires of the 2 Months Post-intervention evaluation but did not complete the remote assessment in which the FMA was administered.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Stroke Survivor | Control Stroke Survivors
Number analyzed (Participants) | 16 | 6
score on a scale
  Baseline | 46.8 (12.2) | 49.0 (10.0)
  2 Months Post-intervention | 50.7 (8.4) | 55.3 (6.0)

15. Secondary Outcome: Neuro-QoL Short Form v1.1 - Satisfaction With Social Roles and Activities Score Among Stroke Survivors
Description: Stroke survivor quality of life and social participation was assessed by the Neuro-QoL Short Form v1.1 - Satisfaction with Social Roles and Activities. This is an 8- item, Likert-type scale about satisfaction in the last 7 days. Neuro-QoL scores are presented as T-scores with a mean of 50 and standard deviation of 10. Scores below 50 indicate below average satisfaction with social roles and activities. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Stroke Survivor | Control Stroke Survivors
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 44.2 (3.4) | 43.2 (4.8)
  2 Months Post-intervention | 45.6 (4.8) | 45.0 (7.7)

16. Secondary Outcome: Caregiver Patient-Reported Outcomes Measurement Information System (PROMIS) Depression - Short Form 6a Score
Description: Depressive symptoms among caregivers was assessed with the 6-item PROMIS Depression - Short Form 6a instrument. Responses are given on a scale from 1 to 5 where 1 = never and 5 = always. Total scores range from 6 to 30 where higher scores indicate greater feelings of depression. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Carepartner | Control Carepartners
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 9.1 (3.9) | 9.5 (2.9)
  2 Months Post-intervention | 8.6 (3.8) | 9.0 (2.3)

17. Secondary Outcome: Neuro-QOL SF v1.0 - Upper Extremity Function (Fine Motor, ADL) Score
Description: Fine motor skills and activities of daily living (ADL) related to upper extremity function was assessed by Neuro-QOL SF v1.0 - Upper Extremity Function (Fine Motor, ADL). This is an 8-item, Likert-type scale assessing the respondent's ability to perform various manual activities of daily life. Responses are given on a 5-point scale where 1 = not at all and 5 = very much. The Neuro-QoL scores are standardized as T-scores with a mean of 50 and standard deviation of 10. Scores below 50 indicate below average upper extremity function. Unadjusted means are presented here.
Time Frame: Baseline, 2 months post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Stroke Survivor | Control Stroke Survivors
Number analyzed (Participants) | 17 | 6
score on a scale
  Baseline | 29.6 (6.7) | 32.8 (13.6)
  2 Months Post-intervention | 35.4 (7.7) | 33.6 (11.7)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning when the study intervention began through the final study assessment at 2 months post-intervention.
Arm/Group | CARE-CITE Carepartner | Control Carepartners | CARE-CITE Stroke Survivor | Control Stroke Survivors
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/6 | 0/17 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/6 | 2/17 | 0/6
Other Adverse Events (participants affected / at risk) | 0/17 | 0/6 | 2/17 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CARE-CITE Carepartner (N=17) | Control Carepartners (N=6) | CARE-CITE Stroke Survivor (N=17) | Control Stroke Survivors (N=6)
Fall requiring hospitalization (unrelated to study intervention) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stroke (unrelated to study intervention) (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CARE-CITE Carepartner (N=17) | Control Carepartners (N=6) | CARE-CITE Stroke Survivor (N=17) | Control Stroke Survivors (N=6)
Fall without injury (unrelated to study intervention) (General disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT04040751/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT04040751/ICF_000.pdf